CLINICAL TRIAL: NCT05152056
Title: Role of MRI and Fine Needle Aspiration in the Diagnosis of Parotid Tumors
Brief Title: MRI and Fine Needle Aspiration in the Diagnosis of Parotid Tumors
Acronym: Parotid
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8454
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Parotid Tumor
Keywords: Parotid Tumor; Diffusion MRI; Perfusion MRI; Aspiration cytology; Fine-needle biopsy
MeSH Terms: conditions — Parotid Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
What value is given to MRI diffusion and perfusion sequences in the diagnosis of parotid tumors? Is a fine needle aspiration associated with MRI systematically necessary? The aim of the research is to study the performance of diffusion and perfusion MRI sequences in the diagnosis of parotid tumors on a large series of cases.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Minor subject (<18 years old)
* Operated for a parotid tumor at Strasbourg University Hospital between January 2009 and June 2020
* Having had in the preoperative assessment an MRI of the parotid, also carried out at the Strasbourg University Hospital.
* Subject (and / or his parental authority) not having expressed, after being informed, his opposition to the reuse of his data for the purposes of this research.

Exclusion criteria:

* Subject (or his parents) who expressed his (their) opposition to participating in the study
* Lack of pathological or MRi results
* Subject under guardianship, curatorship or safeguard of justice

Min Age: 6 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Minor and major subjects operated for a parotid tumor at Strasbourg University Hospital between January 2009 and June 2020 and having had in the preoperative assessment an MRI of the parotid, also carried out at the Strasbourg University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Study the performance of diffusion and perfusion MRI sequences in the diagnosis of parotid tumors on a large series of cases | Files analysed retrospectively from January 1, 2009 to June 30, 2020 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ORL et de Chirurgie Cervico-Faciale - Hôpitaux Universitaires de Strasbourg, Strasbourg, France